CLINICAL TRIAL: NCT00233194
Title: Identification of Sleep-Disordered Breathing in Children
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ronald D. Chervin, M.D., M.S., Michael S Aldrich Collegiate Professor of Sleep Medicine and Professor of Neurology, University of Michigan
Other Study IDs: 324; R01HL080941 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Sleep; Sleep Apnea Syndromes; Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 2: Children scheduled for adenotonsillectomy and healthy subjects, for comparison, not scheduled for such surgery.
  Interventions: Procedure: Observational follow-up study of adenotonsillectomy

INTERVENTIONS:
Procedure: Observational follow-up study of adenotonsillectomy — Studies of sleep, behavior, cognition, and daytime sleepiness
  Other Names: Adenotonsillectomy vs. non-surgical subjects

SUMMARY:
The purpose of this research is to study and improve the methods used to detect childhood breathing problems during sleep that can affect daytime behavior at home and school. Early diagnosis of these sleep disorders may allow doctors to treat children at a time when the consequences can still be reversed.

DETAILED DESCRIPTION:
BACKGROUND:

Sleep-disordered breathing (SDB) affects at least 1 to 3 percent of children. Associated morbidity can include inattentive and hyperactive behavior, disruptive behavior disorders, cognitive deficits, and excessive daytime sleepiness. Sleep specialists recommend that children undergo polysomnography to confirm SDB, especially before undergoing treatment, which often involves an adenotonsillectomy. Unfortunately, such testing is rarely performed either before or after surgery. Available data suggest that a clinical diagnosis of SDB does not predict polysomnographic results reliably. However, the extent to which polysomnographic results predict morbidity, and especially treatable morbidity, is not well known. The main goal of the proposed research, therefore, is to study and improve methods for identification of childhood SDB that carries reversible morbidity.

DESIGN NARRATIVE:

Researchers will examine the utility of polysomnography in a group of children scheduled to undergo adenotonsillectomy for clinical indications, and a group of matched control subjects. Initial evaluations, before surgery in the first group, will be compared to results of identical evaluations 6 months later in this controlled nonrandomized trial. Outcomes will be provided by well-validated assessments of behavior, psychiatric status, cognition, and sleepiness. Explanatory variables will include standard clinical and polysomnographic information, and data from two newer techniques. The first, nasal pressure monitoring, shows increased sensitivity for events that characterize SDB, but few results and no outcome data have been reported from use of this method in children. The second is an innovative signal processing algorithm developed by the investigators to show that cortical electroencephalogram (EEG) activity changes in synchrony with non-apneic respiratory cycles in children with SDB. Preliminary data suggest that the magnitude of respiratory cycle-related EEG changes (RCREC) varies with SDB severity, diminishes after SDB treatment, and improves prediction of neurobehavioral outcomes. The specific aims of the proposed research are to show that 1) nasal pressure monitoring, in comparison to standard measures of airflow, improves prediction of neurobehavioral response to adenotonsillectomy; 2) RCREC, in comparison to standard visually-scored EEG-based arousals, do likewise; 3) polysomnographic SDB measures, including nasal pressure monitoring and RCREC, add useful information to that derived from office-based assessments; and 4) polysomnography after adenotonsillectomy can identify clinically relevant residual SDB in some children.

ELIGIBILITY:
Inclusion Criteria:

* Assent of child (if over the age of 9 or younger but able to understand the nature of the study)
* At least one parent or guardian must sign an informed consent
* Child must be either a healthy volunteer or scheduled for an adenotonsillectomy for any reason
* Children scheduled for adenotonsillectomies must be referred to the program by a treating otolaryngologist who practices at the University of Michigan or St. Joseph Mercy Hospital in Ann Arbor, Michigan

Exclusion Criteria:

* Mental or physical limitations that would prevent proper interpretation of neurobehavioral tests
* Medical history that could confound interpretation of EEG or behavioral data, including epilepsy, psychiatric diagnoses (other than disruptive behavior disorders), head trauma with loss of consciousness for more than 30 seconds, or chronic medication use (e.g., benzodiazepines, other hypnotics, or antihistamines)
* Current treatment by a physician or past surgical treatment for SDB
* A known medical condition that carries independent high risk of SDB (e.g., Pierre Robin syndrome, Down syndrome, or neuromuscular disorders) or excessive daytime sleepiness (e.g., narcolepsy)
* Inability to schedule polysomnography, a Multiple Sleep Latency Test, and neurobehavioral testing before the surgical date
* Determination by any of the patient's physicians that sleep testing is required before surgery can be scheduled (to avoid the possibility that study enrollment itself could affect ability to complete the study)
* Prior enrollment of a sibling in the study
* Expectation that the child will no longer have convenient access to University of Michigan facilities within 6 months or expectation of further surgery within that period

Additional exclusion criteria for healthy volunteers include:

* Any history of adenoidectomy or tonsillectomy
* Plans for either procedure in the future
* History of habitual snoring
* History of large (uninfected) tonsils
* History of recurrent throat infection that might be grounds for adenotonsillectomy (three episodes in each of 3 years, five episodes in each of 2 years, or seven episodes in one year)

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who are scheduled to undergo adenotonsillectomy for clinical indications, as well as a group of control subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2005-01; Primary Completion 2009-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Overall behavior | Measured for approximately 6 months
Psychiatric status | Measured for approximately 6 months
Cognition | Measured for approximately 6 months
Sleepiness (measured immediately before surgery and 6 months after surgery) | Measured for approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Chervin, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] O'Brien LM, Lucas NH, Felt BT, Hoban TF, Ruzicka DL, Jordan R, Guire K, Chervin RD. Aggressive behavior, bullying, snoring, and sleepiness in schoolchildren. Sleep Med. 2011 Aug;12(7):652-8. doi: 10.1016/j.sleep.2010.11.012. Epub 2011 May 26. PMID 21620766
- [Background] Paruthi S, Chervin RD. Approaches to the assessment of arousals and sleep disturbance in children. Sleep Med. 2010 Aug;11(7):622-7. doi: 10.1016/j.sleep.2009.11.018. PMID 20620104
- [Background] Chervin RD, Fetterolf JL, Ruzicka DL, Thelen BJ, Burns JW. Sleep stage dynamics differ between children with and without obstructive sleep apnea. Sleep. 2009 Oct;32(10):1325-32. doi: 10.1093/sleep/32.10.1325. PMID 19848361
- [Background] Giordani B, Hodges EK, Guire KE, Ruzicka DL, Dillon JE, Weatherly RA, Garetz SL, Chervin RD. Neuropsychological and behavioral functioning in children with and without obstructive sleep apnea referred for tonsillectomy. J Int Neuropsychol Soc. 2008 Jul;14(4):571-81. doi: 10.1017/S1355617708080776. PMID 18577286
- [Background] Lumeng JC, Chervin RD. Epidemiology of pediatric obstructive sleep apnea. Proc Am Thorac Soc. 2008 Feb 15;5(2):242-52. doi: 10.1513/pats.200708-135MG. PMID 18250218
- [Background] Dillon JE, Blunden S, Ruzicka DL, Guire KE, Champine D, Weatherly RA, Hodges EK, Giordani BJ, Chervin RD. DSM-IV diagnoses and obstructive sleep apnea in children before and 1 year after adenotonsillectomy. J Am Acad Child Adolesc Psychiatry. 2007 Nov;46(11):1425-36. doi: 10.1097/chi.0b013e31814b8eb2. PMID 18049292
- [Background] Chervin RD, Weatherly RA, Garetz SL, Ruzicka DL, Giordani BJ, Hodges EK, Dillon JE, Guire KE. Pediatric sleep questionnaire: prediction of sleep apnea and outcomes. Arch Otolaryngol Head Neck Surg. 2007 Mar;133(3):216-22. doi: 10.1001/archotol.133.3.216. PMID 17372077
- [Background] Chervin RD, Weatherly RA, Ruzicka DL, Burns JW, Giordani BJ, Dillon JE, Marcus CL, Garetz SL, Hoban TF, Guire KE. Subjective sleepiness and polysomnographic correlates in children scheduled for adenotonsillectomy vs other surgical care. Sleep. 2006 Apr;29(4):495-503. PMID 16676783
- [Background] Chervin RD, Ruzicka DL, Giordani BJ, Weatherly RA, Dillon JE, Hodges EK, Marcus CL, Guire KE. Sleep-disordered breathing, behavior, and cognition in children before and after adenotonsillectomy. Pediatrics. 2006 Apr;117(4):e769-78. doi: 10.1542/peds.2005-1837. PMID 16585288
- [Background] Chervin RD, Ruzicka DL, Archbold KH, Dillon JE. Snoring predicts hyperactivity four years later. Sleep. 2005 Jul;28(7):885-90. doi: 10.1093/sleep/28.7.885. PMID 16124670
- [Background] Chervin RD, Burns JW, Ruzicka DL. Electroencephalographic changes during respiratory cycles predict sleepiness in sleep apnea. Am J Respir Crit Care Med. 2005 Mar 15;171(6):652-8. doi: 10.1164/rccm.200408-1056OC. Epub 2004 Dec 10. PMID 15591467
- [Background] Weatherly RA, Ruzicka DL, Marriott DJ, Chervin RD. Polysomnography in children scheduled for adenotonsillectomy. Otolaryngol Head Neck Surg. 2004 Nov;131(5):727-31. doi: 10.1016/j.otohns.2004.06.699. PMID 15523455
- [Background] Chervin RD, Burns JW, Subotic NS, Roussi C, Thelen B, Ruzicka DL. Correlates of respiratory cycle-related EEG changes in children with sleep-disordered breathing. Sleep. 2004 Feb 1;27(1):116-21. doi: 10.1093/sleep/27.1.116. PMID 14998247
- [Background] Chervin RD, Burns JW, Subotic NS, Roussi C, Thelen B, Ruzicka DL. Method for detection of respiratory cycle-related EEG changes in sleep-disordered breathing. Sleep. 2004 Feb 1;27(1):110-5. doi: 10.1093/sleep/27.1.110. PMID 14998246
- [Background] Chervin RD, Ruzicka DL, Wiebelhaus JL, Hegeman GL 3rd, Marriott DJ, Marcus CL, Giordani BJ, Weatherly RA, Dillon JE. Tolerance of esophageal pressure monitoring during polysomnography in children. Sleep. 2003 Dec 15;26(8):1022-6. doi: 10.1093/sleep/26.8.1022. PMID 14746385
- [Background] Chervin RD, Dillon JE, Archbold KH, Ruzicka DL. Conduct problems and symptoms of sleep disorders in children. J Am Acad Child Adolesc Psychiatry. 2003 Feb;42(2):201-8. doi: 10.1097/00004583-200302000-00014. PMID 12544180
- [Background] Chervin RD, Archbold KH, Dillon JE, Panahi P, Pituch KJ, Dahl RE, Guilleminault C. Inattention, hyperactivity, and symptoms of sleep-disordered breathing. Pediatrics. 2002 Mar;109(3):449-56. doi: 10.1542/peds.109.3.449. PMID 11875140
- [Result] Chung S, Hodges EK, Ruzicka DL, Hoban TF, Garetz SL, Guire KE, Felt BT, Dillon JE, Chervin RD, Giordani B. Improved behavior after adenotonsillectomy in children with higher and lower IQ. Int J Pediatr Otorhinolaryngol. 2016 Jan;80:21-5. doi: 10.1016/j.ijporl.2015.11.005. Epub 2015 Nov 10. PMID 26746606
- [Result] Chervin RD, Chung S, O'Brien LM, Hoban TF, Garetz SL, Ruzicka DL, Guire KE, Hodges EK, Felt BT, Giordani BJ, Dillon JE. Periodic leg movements during sleep in children scheduled for adenotonsillectomy: frequency, persistence, and impact. Sleep Med. 2014 Nov;15(11):1362-9. doi: 10.1016/j.sleep.2014.05.004. Epub 2014 Jun 6. PMID 25218486
- [Result] Chervin RD, Garetz SL, Ruzicka DL, Hodges EK, Giordani BJ, Dillon JE, Felt BT, Hoban TF, Guire KE, O'Brien LM, Burns JW. Do respiratory cycle-related EEG changes or arousals from sleep predict neurobehavioral deficits and response to adenotonsillectomy in children? J Clin Sleep Med. 2014 Aug 15;10(8):903-11. doi: 10.5664/jcsm.3968. PMID 25126038
- [Result] Chervin RD, Ruzicka DL, Hoban TF, Fetterolf JL, Garetz SL, Guire KE, Dillon JE, Felt BT, Hodges EK, Giordani BJ. Esophageal pressures, polysomnography, and neurobehavioral outcomes of adenotonsillectomy in children. Chest. 2012 Jul;142(1):101-110. doi: 10.1378/chest.11-2456. PMID 22302302